CLINICAL TRIAL: NCT04082390
Title: A Randomized, Double-blind, Placebo-controlled Study Evaluating the Effects of the GOLO for Life System Diet With and Without GOLO Release Supplement on Glycemic Control and Insulin Resistance in Overweight and Obese Subjects With Type 2 Diabetes
Brief Title: Effects of the GOLO for Life System Diet With and Without GOLO Release Supplement on Glycemic Control and Insulin Resistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Golo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOLO 1704
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Drainage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RELEASE Supplement (Experimental)
  Interventions: Dietary Supplement: RELEASE
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: RELEASE — Dietary supplement
  Arms: RELEASE Supplement
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind placebo-controlled study is intended to observe the short-term effects of the GFL System Diet with Release supplement versus GFL System Diet with placebo on glycemic metabolism and insulin resistance in patients with Type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years
* Body mass index (BMI) ≥ 27 and ≤ 60 kg/m2
* Have the ability to engage in at least 15 minutes of moderate physical activity such as brisk walking
* A1C greater than or equal to 6.5% at screening
* Willing to comply with study procedures described herein

Exclusion Criteria:

* Current diagnosis of type 1 diabetes
* Subjects with a history of hypoglycemia
* A history of an eating disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Known allergy to any of the components in the Release supplement
* A history of prior surgery for weight loss within one year from screening
* Currently taking injectable medications to control diabetes, including insulin and GLP-1 agonists
* Currently pregnant or breastfeeding or have had a baby within the last six weeks
* Planning to become pregnant in the next three months. Women of child-bearing potential must be willing and able to use adequate and reliable contraception throughout the study (e.g. abstinence or barrier with additional spermicidal foam or jelly, or the use of intrauterine device or hormonal contraception).
* Uncontrolled hypertension at screening defined as Systolic blood pressure greater than 180 mmHG or Diastolic blood pressure greater than 110 mmHG
* Current clinical diagnosis or signs and symptoms of unstable (in the opinion of the principle investigator) heart, kidney or liver disease, cancer, or chronic neurological disease.
* Current participation in any other weight loss or weight management program
* Currently taking weight loss medications, or medications or supplements known to be associated with significant weight loss or weight gain
* Has any condition that, in the opinion of the investigator, would make participation in this study not in the best interest of the subject or that could prevent, limit or confound the protocol-specified assessments. Examples include: history of diabetic ketoacidosis; active chronic liver disease or cirrhosis; chronic autoimmune disease; inflammatory bowel disease, colonic ulceration, partial intestinal obstruction, subjects predisposed to intestinal obstruction; chronic intestinal diseases associated with marked disorders of digestion or absorption

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fasting Blood Glucose (FBG) at approximately 4 weeks of the GFL System Diet with Release supplement versus GFL System Diet with placebo supplement | 4 weeks

SECONDARY OUTCOMES:
Change from baseline in Fructosamine between the 2 groups | 4 weeks
Change from baseline in HGB A1C between the 2 groups | 4 weeks
Change from baseline in Insulin Levels between the 2 groups | 4 weeks
Change from baseline in HOMA-IR between the 2 groups | 4 weeks
Change from baseline in Weight between the 2 groups | 4 weeks
Change from baseline in Body Mass Index between the 2 groups | 4 weeks
Change from baseline in Hip Circumference between the 2 groups | 4 weeks
Change from baseline in Waist Circumference between the 2 groups | 4 weeks
Change from baseline in Blood Pressure between the 2 groups | 4 weeks
Change from baseline in Heart Rate between the 2 groups | 4 weeks

IPD SHARING:
Plan to Share IPD: Undecided